CLINICAL TRIAL: NCT03778437
Title: Aiming Method May Facilitate Needle Alignment in Ultrasound-guided Subclavian Vein Catheterization
Brief Title: Facilitating Needle Alignment With Aiming Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Qingxiang Mao, Principal Investigator, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018(45)
Record Dates: First submitted 2018-12-03; First posted 2018-12-19 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Central Venous Catheters

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- landmark techniques (Active Comparator): Subclavian vein catheterization is performed without the guidance of ultrasound. The needle was inserted 1 cm inferior and 1 cm lateral to the junction of the middle and medial thirds of the clavicle (infraclavicular approach)
  Interventions: Procedure: landmark techniques
- ultrasound-guided with aiming method (Experimental): Subclavian vein catheterization is performed with our newly proposed aiming method with the guidance of ultrasound.
  Interventions: Procedure: subclavian vein catheterization
- ultrasound-guided plus needle guide techniques (Experimental): Subclavian vein catheterization is performed under ultrasound guidance with in-plane technique.
  Interventions: Procedure: Ultrasound-guided plus needle guide techniques

INTERVENTIONS:
Procedure: subclavian vein catheterization — Here we introduced a new freehand method, named as Aiming Method, which facilitated the alignment of injection needles with ultrasound beams. During this aiming method, patient is still positioned in Tredelenburg with the arm abducted to 90° and no needle guidance will be used.
  Arms: ultrasound-guided with aiming method
Procedure: landmark techniques — The patient is positioned in Tredelenburg with the arm abducted to 90°. Venipuncture should occur 1 cm lateral to the curvature of the middle third of the clavicle with the needle pointing horizontally directed at the sternal notch. If subclavian vein is missing at the first try, withdraw the needle and direct horizontally at the cricoid cartilage at the second try.
  Arms: landmark techniques
Procedure: Ultrasound-guided plus needle guide techniques — Subclavian vein catheterization is performed under ultrasound guidance with in-plane technique. The patient is positioned in Tredelenburg with the arm abducted to 90°. During the needle insertion, the needle is secured in the needle guidance device which keeps the alignment of needle and ultrasonic beam.
  Arms: ultrasound-guided plus needle guide techniques

SUMMARY:
Although ultrasound-guided catheterization of the subclavian vein is becoming standard procedure in anesthetic practice, failure to align the needle and the transducer still can lead to possibly complications. In this study, we proposed a new alignment method, namely Aiming Method. The purpose of this study is to investigate whether the use of this aiming method improved resident volunteers' performance of ultrasound-guided SC insertion in real patients. Specifically, residents were asked to perform three different methods: landmark techniques, ultrasound-guided with aiming method and ultrasound-guided plus needle guide techniques.

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 70 years
* American Society of Anesthesiologists (ASA) Physical Status Ⅰ-Ⅲ
* Elective surgery patients requiring subclavian vein catheterization

Exclusion Criteria:

* Local anatomic abnormalities in subclavicular area
* Preexisting subclavian vein thrombosis or coagulation disorders
* Refusal of subclavian vein catheterization

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-27 (Actual)

PRIMARY OUTCOMES:
Procedural time | 24 hours
  the time from skin break to guide wire was positioned into the subclavian vein
Number of skin breaks | 24 hours
  number of skin punctures

SECONDARY OUTCOMES:
The incidence of arterial puncture | 24 hours
  aspiration of arterial blood during needle insertion or local haematoma in ultrasound image
The incidence of pneumothorax | 24 hours
  aspiration of air during needle insertion, or thoracic ultrasonography, or chest radiography

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital, Chongqing, China